CLINICAL TRIAL: NCT02656199
Title: Can the Diaphragm Predict the Course of Mechanical Ventilation? A Prospective Study Evaluating Several M-Mode Ultrasound Measured Diaphragmatic Parameters and Their Effects on Weaning From Mechanical Ventilation
Brief Title: Change In Diaphragmatic Thickness Predicts Extubation Success
Status: Terminated | Type: Observational
Why Stopped: IRB approval expired
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Sponsor
Other Study IDs: 4541
Record Dates: First submitted 2016-01-13; First posted 2016-01-14 (Estimated); Results first posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2016-01

CONDITIONS: Mechanical Ventilation Complication
Keywords: Diaphragm; Ventilators, Mechanical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Main Cohort: all patients enrolled will have an ultrasound of their diaphragm performed once they are on a pressure support trial. Intervention: Diaphragm Ultrasound
  Interventions: Procedure: Diaphragm Ultrasound

INTERVENTIONS:
Procedure: Diaphragm Ultrasound — Once on a pressure support weaning trial, enrolled subjects will have an ultrasound of their right hemidiaphragm performed on three levels of pressure support: 15/5 10/5 and 5/5

SUMMARY:
We will investigate whether measurement of the change in thickness of the diaphragm during the respiratory cycle by ultrasound can predict extubation success in a 48 hour window. We will also asses whether this is only possible on low levels of pressure support as has been shown previously, or if this technique retains its predictive power at higher levels of pressure support.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18, ventilated for >24 hours

Exclusion Criteria:

* already chronically on mechanical ventilatory support, already has tracheostomy, has pathology that obscures visualization of the right hemidiaphragm, has acute stroke either hemorrhagic or ischemic, cannot identify appropriate decision maker to get informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on mechanical ventilation in the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01-13 (Actual); Study Completion 2017-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Blumhof, DO, Principal Investigator — Einstein Healthcare Network
Locations (1):
- Einstein Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 0 participants analyzed. PI has left the institution. Efforts made to contact the PI were unsuccessful. No study data available.
Pre-assignment Details: 0 participants analyzed. PI has left the institution. Efforts made to contact the PI were unsuccessful. No study data available.
Groups:
- Main Cohort: all patients enrolled will have an ultrasound of their diaphragm performed once they are on a pressure support trial. Intervention: Diaphragm Ultrasound
  Diaphragm Ultrasound: Once on a pressure support weaning trial, enrolled subjects will have an ultrasound of their right hemidiaphragm performed on three levels of pressure support: 15/5 10/5 and 5/5
  0 participants analyzed. PI has left the institution. Efforts made to contact the PI were unsuccessful. No study data available.
  PI has left the institution. Efforts made to contact the PI were unsuccessful. No study data available.
Period: Overall Study
Arm/Group | Main Cohort
Started | 0 (0 analyzed.PI left the institution.Effort to contact PI unsuccessful.No study data available)
Completed | 0 (0 analyzed.PI left the institution.Effort to contact PI unsuccessful.No study data available)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: PI has left the institution. Efforts made to contact the PI were unsuccessful. No study data available.
Groups:
- Main Cohort: all patients enrolled will have an ultrasound of their diaphragm performed once they are on a pressure support trial. Intervention: Diaphragm Ultrasound
  Diaphragm Ultrasound: Once on a pressure support weaning trial, enrolled subjects will have an ultrasound of their right hemidiaphragm performed on three levels of pressure support: 15/5 10/5 and 5/5
  PI has left the institution. Efforts made to contact the PI were unsuccessful. No study data available.
Arm/Group | Main Cohort
Number analyzed (Participants) | 0
Age, Categorical — PI has left the institution. Efforts made to contact the PI were unsuccessful. No study data available.
Age, Continuous [unit: PI has left the institution. Efforts mad]
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Extubation Success
Description: Discontinuation from mechanical ventilation in 48 hours from ultrasound
  PI has left the institution. Efforts made to contact the PI were unsuccessful. No study data available.
Time Frame: 48 hours
Population: PI has left the institution. Efforts made to contact the PI were unsuccessful. No study data available.
Arm/Group | Main Cohort
Number analyzed (Participants) | 0

2. Secondary Outcome: Re-intubation
Description: Reinstitution of mechanical ventilation within 48 hours of extubation PI has left the institution. Efforts made to contact the PI were unsuccessful. No study data available.
Time Frame: 48 hours from removal of ventilatory support
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 0 participants analyzed. PI has left the institution. Efforts made to contact the PI were unsuccessful. No study data available.
Description: 0 participant analyzed. PI has left the institution. Efforts made to contact the PI were unsuccessful. No study data available.
Arm/Group | Main Cohort
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
0 Participants analyzed. PI has left the institution. Efforts made to contact the PI were unsuccessful. No study data available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes